CLINICAL TRIAL: NCT07281391
Title: Direct Selective Laser Trabeculoplasty Providing Effective Intraocular Pressure Reduction in Pigmentary Glaucoma Patients
Brief Title: IOP Reduction in Pigmentary Glaucoma Using DSLT
Status: Not yet recruiting | Type: Observational
Sponsor: Mann Eye Institute (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: AH-25-01
Record Dates: First submitted 2025-11-20; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Pigmentary Dispersion Syndrome; Pigmentary Dispersion Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Voyager DSLT — DSLT is an innovative adaptation of traditional SLT. Rather than using a gonioscopic lens, DSLT applies laser energy directly through the limbus to the trabecular meshwork in a few seconds.

SUMMARY:
This study is a single-site, single-arm, prospective, observational study of IOP reduction after DSLT. Subjects will be assessed up to 12 months post-operatively. Clinical evaluations will include IOP and number of glaucoma medications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with pigmentary dispersion syndrome with elevated IOP or mild to moderate (based on AAO Preferred Practice Program criteria) pigmentary glaucoma with glaucomatous optic neuropathy and corresponding visual field/RNFL loss.
* Treatment naive, or washed out IOP ranging from ≥18-34 mmHg
* Central corneal thickness (CCT) 480-600 µm
* Able to complete medication washout and follow-up

Exclusion Criteria:

* Prior incisional glaucoma surgery or glaucoma-related procedures in the study eye
* Prior laser trabeculoplasty <3 years
* Prior intraocular surgery and refractive surgery, except for cataract surgery unless greater than 2 years
* Patients anticipating cataract surgery within the follow-up period
* History of ocular inflammation and infection
* All other secondary glaucoma including exfoliative
* Patients unable to have DSLT treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible test subjects will be adult patients with pigmentary dispersion syndrome with elevated IOP or mild to moderate (based on AAO Preferred Practice Program criteria) pigmentary glaucoma with glaucomatous optic neuropathy and corresponding visual field/RNFL loss.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Mean washed-out IOP change post-DSLT compared to washed-out baseline IOP | 6 months post-DSLT

SECONDARY OUTCOMES:
Complete success: proportion of eyes with ≥ 20% washed out IOP reduction post-DSLT without secondary interventions (additional medications or procedures) compared with washed out baseline IOP | 6 months post-DSLT
Complete success: proportion of eyes with ≥ 20% washed out IOP reduction post-DSLT without secondary interventions (additional medications or procedures) compared with washed out baseline IOP | 12 months post-DSLT
Qualified success: proportion of eyes with IOP reduction (15-20%) without increase in baseline glaucoma medications | 6 months post-DSLT
Qualified success: proportion of eyes with IOP reduction (15-20%) without increase in baseline glaucoma medications | 12 months post-DSLT
Change in number of glaucoma medication(s) | 6 months post-DSLT
  This applies to enrolled eyes already on medications, or to treatment-naive eyes experiencing an increase in medications after DSLT
Change in number of glaucoma medication(s) | 12 months post-DSLT
  This applies to enrolled eyes already on medications, or to treatment-naive eyes experiencing an increase in medications after DSLT
Proportion of medication free eyes post-DSLT | 6 months post-DSLT
  This applies to enrolled eyes already on medications, or to treatment-naive eyes experiencing an increase in medications after DSLT
Proportion of medication free eyes post-DSLT | 12 months post-DSLT
  This applies to enrolled eyes already on medications, or to treatment-naive eyes experiencing an increase in medications after DSLT

CONTACTS AND LOCATIONS:
Overall Officials: Alex Hacopian, MD, Principal Investigator — Mann Eye Institute
Locations (1):
- Mann Eye Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No